CLINICAL TRIAL: NCT00969605
Title: Adaptive Support Ventilation for Faster Weaning in COPD: A Randomized Controlled Trial
Brief Title: Adaptive Support Ventilation in the Weaning of COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Cenk Kirakli,MD, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital, Intensive Care Unit
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IGCEH-ICU-1
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: weaning; adaptive support ventilation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure support ventilation (Active Comparator)
  Interventions: Procedure: Comparison of two different modes for weaning from mechanical ventilation
- Adaptive support ventilation (Active Comparator)
  Interventions: Procedure: Comparison of two different modes for weaning from mechanical ventilation

INTERVENTIONS:
Procedure: Comparison of two different modes for weaning from mechanical ventilation — Chronic obstructive pulmonary disease patients under mechanical ventilation were randomized to adaptive or pressure support ventilation modes when they met the weaning criteria.
  Other Names: weaning protocol

SUMMARY:
Adaptive support ventilation (ASV) is a closed loop ventilation mode that can act both as pressure support (PSV) and pressure controlled (PCV) ventilation. Weaning with ASV shows promising results mainly in post-cardiac surgery patients. The aim of this randomized controlled study was to test the hypothesis that weaning with ASV could reduce the weaning duration in patients with chronic obstructive pulmonary disease (COPD) when compared with PSV.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* On invasive mechanical ventilation for at least 24 hours because of hypoxemic and/or hypercapnic respiratory failure

Exclusion Criteria:

* Mechanical ventilation less then 24 hours (self extubation or death),
* Having a tracheotomy and
* COPD coexisted with severe cardiac or neurologic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Weaning duration

SECONDARY OUTCOMES:
Weaning success
Length of stay in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Kirakli, MD, Study Director — Izmir Dr Suat Seren Chest Diseases and Chest Surgery Education and Research Hospital
Locations (1):
- Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital, Intensive Care Unit, Izmir, Turkey (Türkiye)